CLINICAL TRIAL: NCT02306343
Title: Evaluation of the Effects of Heating the Vicinity of the Insulin Delivery Site by the Experimental Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-148
Record Dates: First submitted 2014-09-03; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus
Keywords: rapid acting insulin; insulin injection; insulin delivery; local heating; experimental device; pre and post meal glucose level
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (with the InsuPad device) (Experimental): In the Meal Tolerance Test protocol - After overnight fast followed by a pre-study stabilization period, the InsuPad device was placed on the abdomen of the subject. The InsuPad device was activated and insulin bolus (0.2 units/kg body weight) was injected right before study start. The injection was given to the subject's abdomen through the injection window of the InsuPad device. Immediately afterwards the subject was asked to drink a standardized liquid meal within 10 minutes. Blood glucose measurements were taken from a peripheral venous line at a pre-determined time points. Total follow up time was 5 hours post meal.
  In the daily life setting - Up to 12 months with the device (test). Subjects were asked to perform at least 3 blood glucose measurements during the day.
  Interventions: Device: InsuPad
- Control (without the InsuPad device) (No Intervention): In the Meal Tolerance Test protocol - After overnight fast followed by a pre-study stabilization period, insulin bolus (0.2 units/kg body weight) was injected to the abdomen right before study start. Immediately afterwards the subject was asked to drink a standardized liquid meal within 10 minutes. Blood glucose measurements were taken from a peripheral venous line at a pre-determined time points. Total follow up time was 5 hours post meal.
  In the daily life setting - Up to 12 months without the device (control). Subjects were asked to perform at least 3 blood glucose measurements during the day.

INTERVENTIONS:
Device: InsuPad — The InsuPad device is composed of a disposable heating pad and a reusable control unit. The heating pad is intended for one day use. The user would attach the InsuPad device to a site where insulin can be injected. When there is a need for insulin bolus injection the user would inject the insulin to a location designate for that. The device would start heating the area around the injection site without over heating the insulin. At the end of the day the subject would remove the device, dispose of the disposable unit and put the reusable unit for recharging.
  Arms: Test (with the InsuPad device)

SUMMARY:
The study is an open-label, randomized, two-period, one-way crossover study using the Meal Tolerance Test (MTT) protocol or the daily life setting protocol.

The study consists of two parts. Subject may participate in both parts or just in one part.

The first part tests the effect of local heating on the post prandial glucose levels following a bolus at in-patient settings.Type I and type II diabetic patients on basal bolus insulin therapy admitted after overnight fast for a meal tolerance test. Subjects injected 0.2 units/kg and consumed standardized liquid meal. Blood samples for glucose and insulin measurements was taken from a venous line. The study was conducted twice with (test) and without (control) the use of the InsuPad device.

The second part evaluate the safety and efficacy of the device use at daily life settings. Type I and type II diabetic patients enrolled to the study. They will be required to perform at least 3 self monitored blood glucose (SMBG) measurements. Study length is up to 25 months. Up to one month run in period, up to 12 months with the device (test) and up to 12 months without the device (control).The subjects will be asked to record events of hypoglycemia, hyperglycemia and any adverse events related to diabetes or the study.

DETAILED DESCRIPTION:
The effect of the InsuPad device was studied using the Meal Tolerance Test protocol or the daily life setting protocol. In the Meal Tolerance Test protocol subjects consumed a standardized liquid meal taken immediately after injection of insulin bolus (0.2 units/kg body weight). Each subject went through the same Meal Tolerance Test protocol twice, once with the InsuPad device (test conditions) and again without the InsuPad device (control conditions) in randomized order. The study started after an overnight fast and stabilization period in which the subject glucose level was stabilized between 100-150 mg/dl, using I.V glucose solution/oral glucose or intravenous insulin administration if needed. The patient remained stable (change of glucose level <20mg/dl) without any intervention or infusion 30 min prior to the study. Blood glucose measurements were taken from a peripheral venous at pre-specified time points. Total follow up time was 5 hours post meal. Safety limits of the study were 75 mg/dl as the low limit and 300 mg/dl as the high limit. If the subject's blood glucose level was below 75 mg/dl glucose solution was given orally to increase his blood glucose level. If subjects blood glucose was above 300 mg/dl iv insulin was given to reduce blood glucose level.

In the daily life setting protocol subjects meeting the inclusion exclusion criteria enrolled to the study. Study length was up to 25 months. Up to one month run in period, up to 12 months with the device (test) and up to 12 months without the device (control). Subjects were asked to perform at least 3 blood glucose measurements a day. Subjects were asked to fill logbooks with measured blood glucose levels and insulin doses given during the whole study. Subjects were asked to report any adverse event during the study. The subjects received a tutorial about the device usage and the study procedures. The order of the test and control phases was randomly selected.

ELIGIBILITY:
Inclusion Criteria:

* Participant age above 18 (including = 18 years)
* BMI above 18kg/m2
* Insulin dependent diabetes using insulin injections
* Diabetic patients with HbA1c values below 12%
* Participant understands the study requirements and the treatment procedures ,willing to comply with all specified follow-up evaluations and provides written Informed Consent before any study-specific tests or procedures are performed

Exclusion Criteria:

* Pregnancy
* Breast feeding women
* Alcohol addiction
* Had Coronary Artery Bypass Graft, are Post Myocardial Infarction or had active Ischemic heart failure in the last 3 months prior to the study date
* Had cardiovascular accident or transient ischemic accident in the last 12 months prior to the study
* Suffer from uncontrolled Hypertension (blood pressure > 165/90)
* Low blood hemoglobin concentration <9 g/dL for female and <12g/dL for male)
* Low Hematocrit concentration <36%; Abnormal kidney and/ or liver function tests. (Creatinine >2 , liver test> 3 times the upper limit of the normal range)
* Psychological incompetence; Any other clinical condition or history, that seems to be relevant to the principle investigator to disqualify the participant
* Subjects with diminished skin integrity
* Subjects with heat sensitivity
* Subjects involved in or planned to participate in other studies that may interfere in data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Blood glucose level during 120 minutes after meal start | 0-120 minutes
  The primary efficacy endpoint of the Meal Tolerance Test (MTT) protocol and of the daily life setting protocol was blood glucose excursion during the first 120 minutes after meal.
Count of mild hypoglycemic events (blood glucose<75) | 5 hours in the Meal Tolerance Test (MTT) protocol and up to 24 months during the daily life setting protocol
  The primary safety endpoint was assessment of the safety of using the InsuPad device including mild hypoglycemia (blood glucose<75).
assessment of skin inflammation | 5 hours in the Meal Tolerance Test (MTT) protocol and up to 24 months during the daily life setting protocol
  The primary safety endpoint was assessment of the safety of using the InsuPad device including skin inflammation.
Count of hyperglycemia events (blood glucose>300) | 5 hours in the Meal Tolerance Test (MTT) protocol and up to 24 months during the daily life setting protocol
  The primary safety endpoint was assessment of the safety of using the InsuPad device including hyperglycemia (blood glucose>300).
assessment of skin irritation | 5 hours in the Meal Tolerance Test (MTT) protocol and up to 24 months during the daily life setting protocol
  The primary safety endpoint was assessment of the safety of using the InsuPad device including skin irritation.

SECONDARY OUTCOMES:
post meal maximal glucose level | 5 hours in the Meal Tolerance Test (MTT) protocol and up to 24 months during the daily life setting protocol
  Secondary endpoint included: post meal maximal glucose level during 5 hours post meal.
area under the curve | 5 hours in the Meal Tolerance Test (MTT) protocol and up to 24 months during the daily life setting protocol
  Secondary endpoint included: area under the curve of the postprandial glucose excursion during 5 hours post meal.

CONTACTS AND LOCATIONS:
Locations (1):
- InsuLine Medical, Petah Tikva, Israel